CLINICAL TRIAL: NCT00205140
Title: Participant Characteristics, Medication Utilization, and the Effects of Pharmacist Initiated Recommendations On the Prescribing For Participants In the Senior MEDS Personalized Medication Review for Adults Age 55 and Older
Brief Title: Effect of Pharmacist Initiated Recommendations On Prescribing For Participants In the Senior MEDS Personalized Medication Review
Status: Terminated | Type: Observational
Why Stopped: The program responsible for recruitment was dismantled in 2006.
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: M-2005-1166
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2015-10

CONDITIONS: Healthy

SUMMARY:
What are the demographic and medication utilization characteristics of participants in the Senior MEDS personalized medication review compared to other community-dwelling elderly, what is the level of satisfaction with Senior Meds, and does the Senior Meds program lead to changes in the participants' drug regimen?

ELIGIBILITY:
Inclusion Criteria:

* 55 or older

Exclusion Criteria:

* 54 or younger

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2005-07; Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Breslow, RPh, BCPS, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States